CLINICAL TRIAL: NCT03266900
Title: A Pilot, Single-centre, Randomized, 5-year, Parallel-group, Superiority Trial to Compare Re-resection of High-grade T1 Bladder Urothelial Carcinoma to no Re-resection for Improving Progression Free Survival
Brief Title: A Superiority Trial to Compare Re-resection of High-grade T1 Bladder Urothelial Carcinoma to no Re-resection for Improving Progression Free Survival
Acronym: RESECT
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulties with accrual
Sponsor: University Health Network, Toronto (Other)
Collaborators: Bladder Cancer Canada (Unknown); Canadian Urological Association (Industry); Canadian Urologic Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-5305.0
Record Dates: First submitted 2017-08-09; First posted 2017-08-30 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Bladder Cancer; Bladder Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- re-TURBT (Experimental): Patients in this arm will receive a 2nd TURBT within 4-6 weeks of initial TURBT
  Interventions: Procedure: re-TURBT
- 6 BCG instillations (Active Comparator): Patients in this arm will not receive a 2nd TURBT, but will receive 6 instillations of BCG.
  Interventions: Drug: 6 weeks BCG instillation

INTERVENTIONS:
Procedure: re-TURBT — 2nd bladder biopsy within 4-6 weeks of initial biopsy
  Arms: re-TURBT
Drug: 6 weeks BCG instillation — standard 6 weeks of BCG induction
  Arms: 6 BCG instillations

SUMMARY:
The investigators would like to compare the progression free survival, overall survival, quality of life, and safety outcomes of patients receiving versus not receiving a 2nd transurethral resection of bladder tumor.

DETAILED DESCRIPTION:
Background: Bladder cancer (BCa) is the 4th and 12th most common malignancies by incidence in Canadian men and women, respectively. In Canada, the lifetime probability of developing BCa is 1 in 27 men and 1 in 84 women. Urologists use a transurethral resection of bladder tumor (TURBT) to diagnose and stage patients with non-muscle invasive bladder cancer (NMIBC). While the value of repeat TURBT is not questioned for incomplete endoscopic resections, retrospective studies have suggested value in repeat resection for high grade T1 (T1HG) tumors even if they are completely resected, typically done within 6 weeks of the initial resection. Repeat TURBT for T1HG BCa has been touted to detect understaged tumors, remove occult residual disease, provide prognostic value and improve subsequent bladder therapy. To date, there is a paucity of high quality level-1 evidence validating repeat TURBT for T1HG compared to a single TURBT for improved long term disease specific outcomes.

Research Question: Among patients with T1HG BCa with completely resected tumor, is repeat TURBT superior to single TURBT for improving 53-year progression free survival (PFS), defined as >/=T2 local disease or lymph node disease/distant metastasis? Study Design: The RESECT trial is designed as a pilot, single-centre, 2-arm parallel-group, superiority randomized trial, with random permuted blocks (lengths of 4 or 6) and balanced allocation (1:1), conducted at the University Health Network.

Patient Population: Adult patients with completely resected T1HG bladder urothelial carcinoma are eligible to participate. Patients with either lymph node/distant metastases at presentation, variant histology, those that had their initial resection performed outside of a study centre, or patients with severe comorbidities are excluded.

Intervention: Repeat TURBT (experimental) versus T1HG standard of care (active control).

Outcomes: The primary outcome is the difference between the two intervention arms with regards to PFS over 5-years of follow-up. Secondary outcomes are the difference between the two intervention arms in: (i) clinical measures; (ii) survival measures; (iii) perioperative safety measures; and (iv) quality of life (QOL) questionnaires.

Randomization: Randomization will occur at the central coordinating site using a computer-generated randomization schedule and random permuted blocks (of lengths 4 or 6). The allocation sequence will be implemented using sequentially numbered, opaque, sealed envelopes.

Blinding: Neither participants nor treating physicians will be blinded to treatment allocation. The research/data analyst team will be blinded as will the radiologists that assess surveillance imaging.

Sample Size: To test feasibility, a sample of 18 cases in 1 year is expected. Analysis: Proportional outcomes will be analyzed with Chi-square or Fisher's exact test and continuous variables will be analyzed with Student's t-test. Time to event outcomes will be analyzed using log-rank tests on Kaplan-Meier estimates, followed by adjusted Cox proportional-hazard models. Continuous variables with differences between two time periods will be analyzed suing an analysis of covariance, with baseline values and centre adjusted for as covariates. Continuous variable outcomes with values over multiple time periods will be analyzed using repeated measures analysis of covariance.

Follow-Up: In addition to baseline assessment, each participant will be followed up at 3, 6, 9, 12, 15, 18, 21, 24, 30, 36, 48, 60 months after the intervention with cystoscopic evaluation, and assessment of disease progression and QOL. Surveillance imaging will be every 6 months for the 5-year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Complete initial resection by a BCa-focused urologic oncologist; mandatory bladder detrusor muscle in the initial TURBT specimen and complete visible resection documented by the surgeon/OR staff by intra-operative photography.
* Urothelial carcinoma as the predominant histology as determined by genitourinary specific pathologist (e.g. small (<50%) components of small cell, squamous cell or adenocarcinoma are allowable).
* Able and willing to consent.
* ≥18 years old: BCa is primarily a disease of the elderly, thus we have elected to include healthy octogenarian/nonagenarian patients. Additionally, since a TURBT can be performed under general or spinal anesthesia, we feel that including these patients is acceptable.

Exclusion Criteria:

* Lymph node or distant metastases at initial presentation - determined on standard BCa staging evaluation with a CT-urogram of the abdomen/pelvis and/or a preoperative chest x-ray demonstrating pulmonary metastases.
* Extensive NMIBC disease warranting immediate cystectomy.
* Variant histology (not urothelial carcinoma) - ie. micropapillary, plasmacytoid, nested or sarcomatoid variants.
* No muscularis propria (inadequate bladder staging) present in the initial TURBT specimen.
* Initial TURBT demonstrating T1HG disease performed outside of study centre - as per study protocol, quality control of surgical performance for this trial requires the TURBT to be performed by an experienced BCa-dedicated surgeon.
* Patients with severe comorbidities, including but not limited to: (i) previous stroke with persistent cognitive, motor, etc deficits; (ii) recent (<6 months) myocardial infarction or current unstable angina; (iii) liver cirrhosis; (iv) severe chronic obstructive pulmonary disease (COPD)/respiratory disease. Patients must be suitable candidates for either spinal or general anesthesia.
* Pregnancy or lactation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2021-10-04 (Actual); Study Completion 2021-10-04 (Actual)

PRIMARY OUTCOMES:
5 year Progression Free Survival | 5 years

SECONDARY OUTCOMES:
Clinical Measures - These include recurrence free survival (in the bladder), time to cystectomy, and metastases-free survival as measured over time from intervention to 5-years post-intervention. | 5 years
  1. Time to bladder recurrence (ie. BCG failure), measured over time from intervention to 5-years post-intervention.
  2. Time to cystectomy, measured over time from intervention to 5-years post-intervention.
  3. Time to metastasis (lymph node or distant metastasis), measured over time from intervention to 5-years post-intervention.
Survival Measures - These include disease specific survival and overall survival as measured over time from intervention to 5-years post-intervention. | 5 years
  1. Time to bladder cancer-specific mortality, measured over time from intervention to 5-years post-intervention
  2. Time to death (examining overall survival), measured over time from intervention to 5-years post-intervention.
Perioperative Safety Measures - These include rate of major complications as defined by the Clavien-Dindo classification as grade 3, 4, and 5. | 5 years
  Proportion with major complications, indicated by the Clavien-Dindo classification of grade 3, 4, and 5, measured during the repeat TURBT hospitalization period.
Mean Change of Patient FACT BI Scores - This includes prospective collection with a validated BCa HRQOL instruments performed at each patient visit. | 5 years
  1. 1-year post-intervention from baseline
  2. Over time at each 3-month surveillance visit (during the first 2 years), each 6-month surveillance visit (during the year 2-3), and each annual surveillance visit (during year 4-5).
  The FACT-Bl metric is validated for measuring HRQOL of patients with BCa. This questionnaire is designed for patients with bladder cancer and includes assessment of four general domains (physical, social/family, emotional and function), with patients responding to statements on a five-point ordinal Likert scale ranging from zero to four. Additionally, there are statements concerning urinary tract symptoms, intestinal symptoms and sexual symptoms (10 statements), with two more for those with a stoma. With 39 statements, the highest score achievable is 156.

CONTACTS AND LOCATIONS:
Overall Officials: Girish Kulkarni, MD PhD FRCSC, Principal Investigator — University Health Network - Princess Margaret Hospital
Locations (1):
- University Health Network, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No